CLINICAL TRIAL: NCT01983644
Title: RECO Flow Restoration Device Versus Solitaire FR With the Intention for Thrombectomy Study: a Prospective Randomised Control Trial(REDIRECT)
Brief Title: RECO Flow Restoration Device Versus Solitaire FR With the Intention for Thrombectomy Study
Acronym: REDIRECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Xinfeng Liu, Professor, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REDIRECT
Record Dates: First submitted 2013-11-04; First posted 2013-11-14 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2016-12

CONDITIONS: Ischemic Stroke
Keywords: acute ischemic stroke,endovascular recanalization; mechanical thrombectomy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RECO thrombectomy (Experimental): IA thrombectomy is executed by RECO flow restoration device which is a novel, self-expanding stent retriever designed to yield rapid flow restoration in acute cerebral ischaemia.
  Interventions: Device: RECO flow restoration device
- Solitaire FR thrombectomy (Active Comparator): IA thrombectomy is executed by Solitaire FR flow restoration device
  Interventions: Device: Solitaire FR flow restoration device

INTERVENTIONS:
Device: RECO flow restoration device — RECO flow restoration device is a novel, self-expanding stent retriever designed to yield rapid flow restoration in acute cerebral ischaemia.
  Other Names: RECO
  Arms: RECO thrombectomy
Device: Solitaire FR flow restoration device — Solitaire FR flow restoration device has been approved by the FDA and CFDA.
  Other Names: Solitaire FR
  Arms: Solitaire FR thrombectomy

SUMMARY:
Endovascular therapy is increasingly used for patients with moderate-to-severe acute ischemic stroke.This study will compare the efficacy and safety of RECO(a novel, self-expanding stent retriever) with Solitaire FR within 8 hours of stroke onset caused by the large vessel occlusion.

DETAILED DESCRIPTION:
RECO is a novel, self-expanding stent retriever, designed to yield rapid flow restoration in acute cerebral ischaemia. The proposed study is a multicenter, randomized, prospective, parallel-group, open-label clinical trial with a blinded outcome, to test the RECO(a novel, self-expanding stent retriever), as compared with Solitaire FR stent retriever.

ELIGIBILITY:
Inclusion Criteria:

1. age (18-80 years)
2. acute ischemic stroke
3. within 8 hours after symptom onset
4. a large-vessel confirmed by CTA/MRA (eg, internal carotid, middle cerebral M1 and/or M2 segments)
5. NIHSS(≥8 and ≤24)
6. patients or their legally authorised representatives provided signed, informed consent.

Exclusion Criteria:

1. CT or MRI evidence of intracranial haemorrhage/tumor
2. major ischaemic infarction (acute ischaemic change in more than a third of the middle cerebral artery territory)
3. NIHSS(≥25 and ≤7)
4. severe sustained hypertension (systolic blood pressure >185 mm Hg or diastolic blood pressure >110 mm Hg)
5. baseline glucose concentrations of less than 2·7 mmol/L or higher than 21.6 mmol/L
6. known haemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with an international normalised ratio of more than 1.7
7. treatment with heparin within 48 h with a partial thromboplastin time more than two times the laboratory normal, baseline platelet count of less than 100×10^9/L
8. history of severe allergy (worse than rash) to contrast medium or nitinol
9. pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2013-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Revascularization Status | Post-procedure, immediate=at the end of the procedure, per last angiogram during treatment
  Revascularization, defined as at least TICI 2a in the vascular territory treated at end of the neuro interventional procedure Thrombolysis in Cerebral Infarction (TICI) grading system for perfusion (ie blood flow through a vessel) Grade 0:No Perfusion. No antegrade flow beyond the point of occlusion. Grade 1:Penetration With Minimal Perfusion. Grade 2:Partial Perfusion. Grade 2a:Only partial filling (<2/3) of the entire vascular territory is visualized. Grade 2b:Complete filling of all of the expected vascular territory is visualized, but slower . Grade 3:Complete Perfusion.

SECONDARY OUTCOMES:
Clinical Outcomes at 90 Days | 90-day
  Good clinical outcome is defined as an modified Rankin Scale (mRS) score of 0-2 at 90 days. mRS 0-2 indicates functional independence 0 - No symptoms.
intracranial hemorrhages | 24 hours
  Incidence of intracranial hemorrhages(ICH) within 24(-6/+12)hours post procedure
all-cause mortality at 90 days | procedure through 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Xinfeng Liu, MD, Study Chair — Department of Neurology, Jinling Hospital, Nanjing 210002, China
Locations (10):
- China (10):
  - Daping Hospital, Chongqing, Chongqing Municipality
  - Fuzhou General Hospital, Fuzhou, Fujian
  - Zhongshan Hospital of Xiamen University, Xiamen, Fujian
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Department of Neurology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Yangzhou First People's Hospital, Yangzhou, Jiangsu
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cao J, Lin H, Lin M, Ke K, Zhang Y, Zhang Y, Zheng W, Chen X, Wang W, Zhang M, Xuan J, Peng Y; REDIRECT Trial Investigators. RECO Flow Restoration Device Versus Solitaire FR With the Intention for Thrombectomy Study (REDIRECT): a prospective randomized controlled trial. J Neurosurg. 2020 Jun 5;134(5):1569-1577. doi: 10.3171/2020.3.JNS193356. Print 2021 May 1. PMID 32502991
- [Derived] Jiang Y, Li Y, Xu X, Yu Y, Liu W, Liu X. An in vitro porcine model evaluating a novel stent retriever for thrombectomy of the common carotid artery. Catheter Cardiovasc Interv. 2016 Feb 15;87(3):457-64. doi: 10.1002/ccd.26285. Epub 2015 Oct 30. PMID 26514251